CLINICAL TRIAL: NCT01390090
Title: Ultrasound Confirmation of Fluoroscopically Guided Piriformis Muscle Injections: Does Accuracy Improve Efficacy?
Brief Title: Ultrasound Confirmation of Fluoroscopically Guided Piriformis Muscle Injections
Status: Withdrawn | Type: Observational
Why Stopped: The Principal Investigator left the University
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 700-2010
Record Dates: First submitted 2011-06-29; First posted 2011-07-08 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Subjects Will Have Failed Conservative Treatment
Keywords: piriformis muscle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects will have failed conservative treatment, including, but not limited to oral medications, physical therapy, manual manipulation, and/or alternative medicine. They will be evaluated by a spine specialist in the Spine Division of the Department of Orthopaedics and will be scheduled for a piriformis muscle (PM) corticosteroid injection.

ELIGIBILITY:
Inclusion Criteria:

* Subject Scheduled to receive piriformis injection for buttock pain
* Baseline pain visual analogue scale (VAS) value of at least 4 on a scale of 0-10 points
* Subjective complaint of pain in the buttocks with radiation down the thigh and/or leg
* Objective clinical diagnosis of piriformis syndrome
* Reproduction of pain with maneuvers that stretch or contract the piriformis muscle over the sciatic nerve

Exclusion Criteria:

* Litigation
* Those receiving long-term (>6 months) remuneration for their pain or seeking new or increased long-term remuneration
* Those unable to read English and complete the assessment instruments
* Diagnosis of systemic inflammatory arthritis (e.g. rheumatoid, lupus)
* Addictive behavior, severe clinical depression or psychotic features. The subjects will be identified at the sole discretion of the PI who per the current standard of care will consent the potential subjects to the study
* Possible pregnancy or other reason that precludes the use of fluoroscopy. Fluoroscopy is the current standard of care for piriformis injections. Its use in this study is no different than the standard of care and will be no different if the subjects are enrolling in the study or not
* Contra-indication to corticosteroid, including known allergies or sensitivities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will have failed conservative treatment, including, but not limited to oral medications, physical therapy, manual manipulation, and/or alternative medicine.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Ultrasound evaluation of fluoroscopically guided needle placement in the piriformis muscle. | Following fluoroscopic guidance of the needle placement and prior to the injection, the needle position will be evaluated by ultrasound.
  Following the fluoroscopically guided needle placement, the non-invasive ultrasound probe will then be placed on the skin with gel and will be used to visualize the needle tip and evaluate the accuracy of the fluoroscopically guided needle placement. Needle placement will be recorded as either inside or outside the piriformis muscle.

CONTACTS AND LOCATIONS:
Overall Officials: D J Kennedy, MD, Principal Investigator — University of Florida